CLINICAL TRIAL: NCT05808634
Title: An Open-label, Multicenter, Phase 1 Study Evaluating the Safety, Pharmacokinetics, and Efficacy of BA3182, a Bispecific Epithelial Cell Adhesion Molecule (EpCAM)/CD3 Antibody, in Patients With Advanced Adenocarcinoma
Brief Title: Phase 1 Study Evaluating BA3182 in Patients With Advanced Adenocarcinoma.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioAtla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA3182-001
Record Dates: First submitted 2023-03-17; First posted 2023-04-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Adenocarcinoma
Keywords: Advanced; Metastatic; Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BA3182 (Experimental): All Patients will receive BA3182
  Interventions: Drug: BA3182

INTERVENTIONS:
Drug: BA3182 — Conditionally active biologic (CAB)-bispecific T-cell engager antibody construct targeting EpCAM

SUMMARY:
The objective of this study is to assess safety and efficacy of BA3182 in Advanced Adenocarcinoma

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase 1 study designed to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of BA3182 in patients with advanced adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced unresectable or metastatic adenocarcinoma
* Age ≥ 18 years
* Adequate renal function
* Adequate liver function
* Adequate hematological function
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Patients must not have clinically significant cardiac disease.
* Patients must not have known non-controlled CNS metastasis.
* Patients must not have active autoimmune disease or a documented history of autoimmune disease.
* Patients must not have a history of ≥ Grade 3 allergic reactions to mAb therapy as wellas known or suspected allergy or intolerance to any agent given during this study.
* Patients must not incomplete recovery from the effects of major surgery or significant traumatic injury before the first dose of study treatment.
* Patients must not have known human immunodeficiency virus (HIV) infection, active hepatitis B and/or hepatitis C.
* Patients must not be women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: Assess dose limiting toxicity as defined in the protocol | Up to 24 months
  Phase 1 Part 1: Safety Profile of BA3182
Part 1: Assess maximum tolerated dose as defined in the protocol | Up to 24 months
  Phase 1 Part 1: Safety Profile of BA3182
Part 2: Confirmed overall response rate (ORR) per RECIST v1.1 | Up to 24 months
  Phase 1 Part 2: Antitumor activity of BA3182

SECONDARY OUTCOMES:
Confirmed overall response rate (ORR) per RECIST v1.1 | Up to 24 months
  Phase 1 Part 1: Antitumor activity of BA3182
Confirmed best overall response best overall response (BOR) | Up to 24 months
  Phase 1: Antitumor activity of BA3182
Confirmed duration of response (DOR) | Up to 24 months
  Phase 1: Antitumor activity of BA3182
Confirmed progression-free survival (PFS) | Up to 24 months
  Phase 1: Antitumor activity of BA3182
Confirmed disease control rate (DCR) | Up to 24 months
  Phase 1: Antitumor activity of BA3182
Confirmed time to response (TTR) | Up to 24 months
  Phase 1: Antitumor activity of BA3182
Confirmed overall survival (OS) | Up to 24 months
  Phase 1: Antitumor activity of BA3182
Confirmed percent change from baseline in target lesion sum of diameters. | Up to 24 months
  Phase 1: Antitumor activity of BA3182
Area under the plasma concentration versus time curve (AUC) | Up to 24 months
  Phase 1: Pharmacokinetics of BA3182
Peak Plasma Concentration (Cmax) Phase 1: Pharmacokinetics | Up to 24 months
  Phase 1: Pharmacokinetics of BA3182
Incidence of anti-drug antibody (ADAs) to BA3182 Phase 1: Pharmacokinetics Phase 1: Immunogenicity | Up to 24 months
  Phase 1: Immunogenicity of BA3182
Incidence of neutralizing antibodies (nAbs) to BA3182. | Up to 24 months
  Phase 1: Immunogenicity of BA3182

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UC Irvine, Irvine, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Fred Hutch Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No